CLINICAL TRIAL: NCT03814863
Title: China Red Eye Study
Acronym: CRES
Status: Completed | Type: Observational
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Xiaofeng Lin, associate dean of Zhongshan Ophthalmic Center, Sun Yat-sen University, Sun Yat-sen University
Other Study IDs: ZOC
Record Dates: First submitted 2018-11-08; First posted 2019-01-24 (Actual); Last update posted 2020-04-14 (Actual); Status verified 2020-04

CONDITIONS: Red Eye
Keywords: red eye; conjunctival congestion; ophthalmology clinic

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No

SUMMARY:
This study intends to use a hospital-based multi-center cross-sectional study to understand the disease composition of "red-eye" patients in Chinese ophthalmology clinics. This study will provide important clinical diagnosis and treatment data for common eye diseases in China with "red eye" as the main performance.

DETAILED DESCRIPTION:
Red eye is a common sign of eye diseases. Eye diseases such as ocular surface inflammation, glaucoma, and uveitis can be expressed as red eyes. The disease with red eye as the main complaint is the most common condition that clinicians need to identify. It is not uncommon to be misdiagnosed and missed clinically. The collection and analysis of the disease composition of the "red eye" in Chinese ophthalmology clinics will help to understand the current status of "red eye" related diseases and provide a systematic and comprehensive clinical basis for the differential diagnosis of red eye.

ELIGIBILITY:
Inclusion Criteria:

* Confirmation of signs under the slit lamp is red eye

Exclusion Criteria:

* The investigator believes that there are any unsuitable reasons for participating in the trial.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with "red eye".
Sampling Method: Non-Probability Sample
Enrollment: 4382 (Actual)
Dates: Start 2018-08-01 (Actual); Primary Completion 2019-12-31 (Actual); Study Completion 2019-12-31 (Actual)

PRIMARY OUTCOMES:
medical diagnosis of each patient | 1 day (when the patient come the the doctor)
  the investigators record patients' diagnosis on questionnaire when the patient come to the doctor

CONTACTS AND LOCATIONS:
Locations (9):
- China (9):
  - Zhongshan Ophthalmic Center of Sun yat-sen Universtiy, Guangzhou, Guangdong
  - Hainan Eye Hospital and Key Laboratory of Ophthalmology, Zhongshan Ophthalmic Center, Sun Yat-sen University, Haikou, Hainan
  - West China Hospital of Sichuan University, Chengdu
  - Affiliated Zhongshan Hospital of Dalian University, Dalian
  - First Affiliated Hospital of Kunming Medical University and Hainan Eye Hospital, Kunming
  - Nanxishan Hospital of Guangxi Zhuang Autonomous Region, Nanning
  - Xin Hua Hospital Affiliated to Shanghai Jiao Tong University School of Medicine, Shanghai
  - llege of Huazhong University of Science and Technology, Wuhan
  - the first affiliated hospital of Xinjiang medical university, Xinjiang